CLINICAL TRIAL: NCT04787653
Title: Evaluation of the OtoBand as a Treatment to Reduce the Perceived Loudness of Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Otolith Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OLith10801
Record Dates: First submitted 2021-02-09; First posted 2021-03-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will be assigned to one of the study's two arms. Participant's in Arm One will receive the effective device first and the placebo device second. Participants in Arm Two will receive the placebo device first and then the effective OtoBand. At the midpoint of a participant's enrollment, the first device will be returned and the second device sent. The participants and researchers will be blinded to which arm of the study a participant is assigned so they will not know if the device in use is effective or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Otoband efficacy on Tinnitus (Active Comparator): Participants will wear the Otoband on the flat part of the right mastoid bone, about an inch behind the pinna and level with the ear canal. Each participant will select his/her preferred stimulation level. The OtoBand will be programmed to operate at one of three power levels that are thought to be effective. The OtoBand will record what power level is selected and how long it was operating at that power level as well as the date and time a usage started. The "use log" will be downloaded at Otolith's lab once the device is received. The participant will wear the device for 30 minutes and record their Tinnitus level in a Google Form.
  Interventions: Device: Otoband
- Placebo device efficacy on Tinnitus (Placebo Comparator): The placebo device will use the same case, headband and battery as the OtoBand. The transducer in the OtoBand will be rotated 90 degrees, so that the placebo device will vibrate in a direction ineffectual at providing bone conducted vibrations. The vibrations will be in the horizontal plane, parallel to the skull, and will not have their energy penetrating the skull all the way to the vestibular system. Each participant will select his/her preferred stimulation level. The placebo devices will be made to vibrate at one of three power levels, none of which are thought to be effective. The placebo will record what power level is selected and how long it was operating at that power level as well as the date and time a usage started. The "use log" will be downloaded at Otolith's lab once the device is received. The participant will wear the device for 30 minutes and record their Tinnitus level in a Google Form.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Otoband — Participants with Tinnitus will wear the Otoband set at an effective power level during a 30 minute time frame and outcome measurements will be recorded in a Google Form.
  Arms: Otoband efficacy on Tinnitus
Device: Placebo — Participants with Tinnitus will wear the Otoband set at a non-effective power level during a 30 minute time frame and outcome measurements will be recorded in a Google Form.
  Arms: Placebo device efficacy on Tinnitus

SUMMARY:
This proposed study is a blinded study in which the participant will wear the OtoBand when their tinnitus is present to determine if the OtoBand reduces the perceived loudness of their tinnitus. The Study will be placebo controlled with each participant using an effective device for half of the enrollment period and a placebo device for half of the enrollment period. The order of placebo and effective usage will be randomized, and the researchers will be blinded to which device a participant is using. Study participants will be instructed in an online telehealth conference on how to operate the OtoBand and how to wear the OtoBand. Participants will be enrolled for approximately 30 days from Informed Consent to Wrap-up call.

DETAILED DESCRIPTION:
This study seeks to gather data on the effect of the OtoBand in participants who have reported symptoms of tinnitus. The study is designed to be conducted remotely using video conferencing between representatives of the manufacturer of the OtoBand and participants. In order to comply with requirements for non-essential contact due to the Covid-19 pandemic, there will be no in-person contact in the study.

Otolith Sound (hereafter: "Otolith") seeks to recruit study participants via several online channels including Facebook, Google and their website https://otolithlabs.com/tinnitustelehealthstudy/ . Otolith will use online advertisements to inform potential participants about the study and ask them to volunteer for online screening and enrollment.

Each participant will be enrolled in the study only after a successful video screening including agreement to participate. After a participant is enrolled, a device will be shipped to them via USPS or similar carrier. The participant will be instructed not to open the shipping box with the device until their initial study call with the study coordinator.

During the initial study call, participants will be instructed on how to use the OtoBand and how to wear the device. There will be a total of four online meetings with each study participant. It is expected that a typical participant will be enrolled in the study for approximately 30 days - from consent to filling out the last questionnaire and online wrap up meeting. In these 30 days, the participant will be wearing a device for 30 minutes each day over the course of two times 5 days. In addition to online study calls, Sponsor will use email and text messaging to communicate with the participants. For example, if a study participant does not complete a study diary on a given day, a text message will be sent reminding them to do so.

After the enrollment period, participants will be instructed to return the device in a pre-paid envelope. The devices will stop functioning 20 days after the first use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 to 70 years old
* Tinnitus that has been present for at least 90 days
* Tinnitus that is constant or predictable
* Computer and access to internet for online video conference
* Score greater than or equal to 36 on the Tinnitus Handicap Questionnaire
* Access to a PayPal, Venmo account to receive compensation

Exclusion Criteria:

* Tinnitus that first presented within the last 90 days
* Tinnitus Handicap Questionnaire of 29 or less
* Skull base surgery within the last 90 days
* Any skull implant (cochlear implant, bone conduction implant, DBS)
* No history of vitreous detachment in the last 60 days (no new floaters or unexplained flashes of light in the eye)
* Taking benzodiazepines (e.g. clonazepam, lorazepam, diazepam) Participant reports that their tinnitus is caused by a medication they are taking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in bothersomeness of Tinnitus as measured by Tinnitus Handicap Questionnaire | Forms filled out daily over two week period by the study participant
  The primary endpoint will be the change in THQ score of a participant while wearing an effective device versus the THQ score at enrollment/baseline.

SECONDARY OUTCOMES:
Change in Quality of Life Measures as measured by the Tinnitus Handicap Questionnaire | Forms filled out daily over two week period by the study participant
  Change in Quality of Life Measures at the conclusion of the study versus the start of enrollment as measured by the Tinnitus Handicap Questionnaire.
Identification of a preferred power level for tinnitus as determined by Otoband device log. | Device use log over two week period of use by the study participant
  Identification of a preferred power level for tinnitus as determined by the power level that participants use for the longest cumulative use throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Principal Investigator — Otolith Labs
Locations (1):
- OtolithLabs https://otolithlabs.com/tinnitustelehealthstudy/, Washington D.C., District of Columbia, United States